CLINICAL TRIAL: NCT00353327
Title: Passive Immunotherapy in HIV-Infected Patients Who Fail to Respond to Multiple Highly Active Antiretroviral Treatment. Randomized Study in Two Phases.
Brief Title: Study of the Effectiveness of Passive Immunotherapy in HIV-Infected Patients Who Are in Virologic Failure
Status: Suspended | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Felipe García, Hospital Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PIT-01
Record Dates: First submitted 2006-07-17; First posted 2006-07-18 (Estimated); Last update posted 2008-03-31 (Estimated); Status verified 2008-03

CONDITIONS: HIV Infection
Keywords: HIV; Passive immunotherapy
MeSH Terms: conditions — HIV Infections

INTERVENTIONS:
Procedure: Plasma infusion

SUMMARY:
To study the effect of passive immunotherapy (PIT) over the HIV-viral load and the CD4 T+-cell counts in patients who have failed to respond to three different Highly-Active Antiretroviral Therapy (HAART), and who have at the moment less than 100 CD4+-T cells/ml and a viral load over 20,000 copies/ml.

DETAILED DESCRIPTION:
Double blind comparative randomized study with placebo in two phases:

Phase I: I: A pilot study to asses the virologic efficacy in 30 patients will be done. They will be under the same HAART regimen, and they will be randomized to receive:

1. Group I: HAART + PIT (n= 15)
2. Group II: HAART + placebo (non-hyperimmune plasma) (n= 15)

Passive immunotherapy will consist in 500 cc of inactivated plasma with methylene-blue (standard inactivation method) from asymptomatic patients in early phases of the infection. A transfusion will be done, and a complete blood test including viral load and CD4+-T cell counts will be done at days 3, 7, 14, 21 and 28. The non-hyperimmune plasma (Group II) will be inactivated by the same method.

A second dose of hyperimmune plasma and placebo (Group I and Group II respectively) will be administered at +1 month from the beginning of the trial.

A complete blood test including viral load and CD4+-T cell counts will be done at month +2, +3 and +4.

Phase II: 30 patients under the same HAART regimen will be randomized to receive:

1. Group I: HAART + PIT (n= 15)
2. Group II: HAART + placebo (non-hyperimmune plasma) (n= 15)

Passive immunotherapy will consist in 500 cc of inactivated plasma with methylene-blue (standard inactivation method) from asymptomatic patients in early phases of the infection, guided by the neutralization capacity of the plasma donors over the virus' receptor . A transfusion will be done, and a complete blood test including viral load and CD4+-T cell counts will be done at days 3, 7, 14, 21 and 28. The non-hyperimmune plasma (Group II) will be inactivated by the same method.

A second dose of hyperimmune plasma and placebo (Group I and Group II respectively) will be administered at +1 month from the beginning of the phase II.

The patients will remain under HAART the next year. A complete clinical examination, and a blood test that includes hemogram and biochemical parameters (renal and hepatic function), and viral load will be done each month. Every three months, a CD4+/CD8+ T cell count will be done, and it will be obtained plasma and serum from each patient.

Additionally, a genotype and a virtual phenotype of the HIV will be obtained at the beginning and at the end of the study.

Study end-points:

-Main end-point: Phase I: proportion of patients who reduce their plasma viral load > or = 1 log after two infusions of hyperimmune plasma.

Phase II: proportion of patients who reduce their plasma viral load > or = 1 log after a year.

- Secondary end-points:

1. Proportion of patients whose CD4+ T cell count is over 100 cells/mm3 after a year.
2. Proportion of patients whose p24-antigenemia is below the limits of detection.
3. Number of mutations conferring resistance to antiretrovirals at the end of the study compared to the mutations at the beginning.
4. Type C events.
5. Death.
6. Toxicity.
7. Adherence.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected patients (CDC C category) confirmed by a Western-blot
* CD4 T cell count under 100/ml form 6 months before the inclusion, and who have never been over 600 CD4 T cells/ml in the last 6 months, even if they have been receiving HAART.
* The patients have received at least 3 different HAART regimens, and they have failed to respond (define failure: CD4 T cell count under 100/ml and plasma viral load over 20,000 copies/ml).
* Plasma viral load over 20,000 copies/ml during at least 6 months.
* Written informed consent
* 18 years old or older

Exclusion Criteria:

* Asymptomatic patients who fill the A category of the CDC (1993)
* Younger than 18 years old
* Who are not expected to accomplish the treatment or the follow up visits
* Pregnancy, breast-feeding women, or women who want to get pregnant
* Denied consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2006-10

PRIMARY OUTCOMES:
Lowering of plasma viral load after the first plasma infusion
Lowering of plasma viral load after a year

SECONDARY OUTCOMES:
Elevation of CD4 T cell count
Negativation of p24 HIV antigen
HIV RNA mutations conferring resistance to HAART
Development of C-events
Dead
Toxicity
Accomplishment

CONTACTS AND LOCATIONS:
Overall Officials: Felipe Garcia, MD, PhD, Principal Investigator — Hospital Clinic of Barcelona
Locations (1):
- Hospital Clínic Barcelona, Barcelona, Spain